CLINICAL TRIAL: NCT02290067
Title: EVALUATING SYSTEM ACCURACY AND USER PERFORMANCE OF BLOOD GLUCOSE MONITORING SYSTEMS FOR SELF-TESTING IN MANAGING DIABETES MELLITUS
Brief Title: System Accuracy and User Performance of Blood Glucose Monitoring Systems for Self-Testing in Managing Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Collaborators: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPM-G-V-1203; IDT-1340-BE (Other: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm)
Record Dates: First submitted 2014-10-22; First posted 2014-11-13 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes
Keywords: blood glucose monitoring system; system accuracy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omnitest 3 (Active Comparator): Blood glucose monitoring system
  Interventions: Device: Blood glucose monitoring system (Omnitest 3)
- Omnitest 5 (Experimental): Blood glucose monitoring system
  Interventions: Device: Blood glucose monitoring system (Omnitest 5)
- Omnitest 5D (Experimental): Blood glucose monitoring system
  Interventions: Device: Blood glucose monitoring system (Omnitest 5D)

INTERVENTIONS:
Device: Blood glucose monitoring system (Omnitest 3)
  Arms: Omnitest 3
Device: Blood glucose monitoring system (Omnitest 5)
  Arms: Omnitest 5
Device: Blood glucose monitoring system (Omnitest 5D)
  Arms: Omnitest 5D

SUMMARY:
The aim of this test is to determine the system accuracy and user performance evaluation of three Blood Glucose Monitoring systems. For system accuracy evaluation the measurement data should cover the whole range of glucose concentration which could usually be expected in patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 1 or type 2 diabetes and healthy subjects
* Signed and dated informed consent form
* For small modifications of the insulin doses to achieve certain blood glucose values (system accuracy evaluation): Male or female subjects with diabetes mellitus type 1 with intensified insulin therapy (intensified conventional therapy) or insulin pump therapy (continuous subcutaneous insulin infusion)

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute illness that in the opinion of the investigating physician might confound the results of the test or which could result in a risk to the patient caused by the test
* Mental incapacity or language barriers precluding adequate compliance with the test procedures
* Severe chronic illness besides diabetes mellitus as assessed by the investigating physician that might confound the results of the test or which could result in a risk to the patient caused by the test
* Legal incompetence or limited legal competence
* Dependency from the sponsor or the clinical investigator (e.g. coworkers of the sponsor or the clinical research center)
* For user performance evaluation: Subjects having used the test systems before themselves or having participated in a study with these Blood Glucose Monitoring Systems
* For system accuracy evaluation: subjects intended to provide blood samples with glucose concentrations between 50 and 80 mg/dl must not have coronary heart disease, myocardial infarction in history, cerebral events in history, peripheral artery occlusive disease- or impaired hypoglycaemia awareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
System accuracy, results obtained from fingertip using blood glucose monitoring systems compared to a reference equipment | up to 6 hours
User performance of blood glucose monitoring systems indicated by patient [questionnaire] | up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nina Jendrike, Dr. med., Principal Investigator — Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft, Ulm, Germany